CLINICAL TRIAL: NCT00549523
Title: A Randomized, Double-blind, Placebo-Controlled Study of the Safety and Efficacy of Lessertia Frutescens (L.)Goldblatt and J.C. Manning (Syn. Sutherlandia Frutescens (L.)R. Br.)in HIV-infected South African Adults
Brief Title: A Controlled Study of the Safety and Efficacy of Lessertia Frutescens in HIV-infected South African Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); Office of Dietary Supplements (ODS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: U19AT003264-01 (NIH); U19AT003264-01 (NIH); TICIPS002_RP01 (E295/05) (Other Grant/Funding Number: Office of Dietary Supplements)
Record Dates: First submitted 2007-10-24; First posted 2007-10-26 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: HIV Infections
Keywords: HIV; Alternative Medicine; Complementary Medicine
MeSH Terms: conditions — HIV Infections | interventions — Contraceptives, Oral

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Placebo (capsule filled with inert materials)
  Interventions: Drug: Placebo
- Low Dose (Experimental): 400 mg bid Lessertia Frutescens
  Interventions: Drug: Low Dose
- Mid Dose (Experimental): 800 mg bid Lessertia Frutescens
  Interventions: Drug: Mid Dose
- High Dose (Experimental): 1200 bid Lessertia Frutescens
  Interventions: Drug: High Dose

INTERVENTIONS:
Drug: Placebo — Capsules containing 0 mg bid (placebo)
  Arms: Placebo
Drug: Low Dose — Capsules containing 400 mg bid of L. frutescens.
  Other Names: Lessertia Frutescens; Sutherlandia
  Arms: Low Dose
Drug: Mid Dose — Capsules containing 800 mg bid of L. frutescens.
  Other Names: Lessertia Frutescens; Sutherlandia
  Arms: Mid Dose
Drug: High Dose — Capsules containing 1200 mg bid of L. frutescens.
  Other Names: Lessertia Frutescens; Sutherlandia
  Arms: High Dose

SUMMARY:
The study is a 2-stage, double-blind, randomized, placebo-controlled study in which fifty-six HIV-positive subjects will be randomized into the first stage. Interim analysis to determine continuation to stage 2 will be performed to determine continuation after 8 subjects per arm have completed a 24-week dosing regimen.

Primary objectives are to determine the safety of Lessertia frutescens when used by HIV-1 infected adults with early disease, and to document the impact of Lessertia frutescens on markers of HIV disease progression. Secondary objective is to determine the effect of Lessertia frutescens on quality of life in HIV-infected adults and length of infection.

DETAILED DESCRIPTION:
The study is a 2-stage, double-blind, randomized, placebo-controlled study following a two-stage, statistical selection theory design. Fifty-six HIV positive subjects will be randomized onto Stage 1 that will comprise a 4-arm parallel group (one placebo and 3 treatment groups) trial. One or possibly two interim analyses will be performed to determine continuation to Stage 2. A blinded interim analysis to determine the superior active treatment arm of Stage 1 will be continued to Stage 2 after 8 subjects per arm have completed the 24-week dosing regimen and the interim analysis. The study will be terminated if the interim analysis identifies either significant safety issues, or demonstrable non-significance. Following a significant outcome in the blinded interim analysis, the selected active and placebo control arms will continue blinded until total n=48 participants per arm for the placebo and selected treatment group have completed 24 weeks per arm. Respective groups will receive capsules containing L. frutescens in dosages of 0 (placebo material), 400mg bid, 800 mg bid or 1200 mg bid in the first stage. Progression to stage 2 will utilize a two arm design in which 34 subjects will receive either 0 mg L. frutescens (placebo) or the active dosage of L. frutescens bid for 24 weeks.

Primary objectives are to determine the safety of Lessertia frutescens when used by HIV-1 infected adults with early disease, and to document the impact of Lessertia frutescens on markers of HIV disease progression. Secondary objective is to determine the effect of Lessertia frutescens on quality of life in HIV-infected adults and length of infection.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 - 65 years
* HIV-1 infection documented by two different rapid tests for HIV-1 antibodies
* CD4 count >350 cells/ul
* Viral load< 20,000 copies/mL
* Normal hematological function
* Absence of clinically significant renal disease
* Normal liver function
* Random glucose < 11.1 mmol/L
* Normal electrocardiogram
* Regular attendance at the Wellness Clinic for at least 4 visits
* Cognitive capacity sufficient to provide informed consent

Exclusion Criteria:

* Any AIDS-defining diagnosis
* Weight loss > 5% of body weight within the preceding six months
* Other features of undiagnosed tuberculosis (including cough, fatigue, drenching night sweats and abnormal chest radiograph)
* Any other significant disease (active TB, hypertension, diabetes mellitus and other endocrine disorders, peptic ulcer disease, gastrointestinal malabsorption, psychiatric illness) either newly diagnosed or controlled by medication.
* Use of any allopathic or traditional medicine other than isoniazid for TB prophylaxis.
* Prior or current use of antiretroviral therapy
* History of allergic conditions or drug allergy/hypersensitivity
* Either history or family history of autoimmune disease
* Alcohol use of >7 units per week or >3 per session, tobacco use of more than 10 cigarettes per day or description of recreational drug use within the past 6 months.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2008-04; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Primary: determine safety of L. frutescens when used by HIV-1 infected adults with early disease, and to document disease progression. | 24 week treatment period

SECONDARY OUTCOMES:
Secondary: Determine the effect of L. frutescens on quality of life in HIV-1 infected adults, and length of infection. | 24 week treatment period

CONTACTS AND LOCATIONS:
Overall Officials: William Folk, Ph.D., Principal Investigator — University of Missouri-Columbia School of Medicine
Locations (1):
- Department of Medicine, Edendale Hospital, Pvt Bag X 509, Pietermaritzburg, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johnson Q, Syce J, Nell H, Rudeen K, Folk WR. A randomized, double-blind, placebo-controlled trial of Lessertia frutescens in healthy adults. PLoS Clin Trials. 2007 Apr 27;2(4):e16. doi: 10.1371/journal.pctr.0020016. PMID 17476314
- [Derived] Wilson D, Goggin K, Williams K, Gerkovich MM, Gqaleni N, Syce J, Bartman P, Johnson Q, Folk WR. Consumption of Sutherlandia frutescens by HIV-Seropositive South African Adults: An Adaptive Double-Blind Randomized Placebo Controlled Trial. PLoS One. 2015 Jul 17;10(7):e0128522. doi: 10.1371/journal.pone.0128522. eCollection 2015. PMID 26186450